CLINICAL TRIAL: NCT05716724
Title: A Prospective, Non-interventional Study, Investigating Glycaemic Control and Treatment Patterns Associated With the Use of Once-daily Oral Semaglutide in Type 2 Diabetes Patients Who Intend to Fast During Ramadan in the United Arab Emirates, Saudi Arabia, and Kuwait
Brief Title: O-SEMA-Fast: A Research Study to Understand How Oral Semaglutide Works in People With Type 2 Diabetes Who Plan to Fast During Ramadan in the United Arab Emirates, Saudi Arabia, and Kuwait
Acronym: O-SEMA-Fast
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN9924-7577; U1111-1280-0404 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-01-29; First posted 2023-02-08 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with T2D: The study is non-interventional as there are no interventions involved and the decision to initiate oral semaglutide treatment is at the discretion of the treating physician and is clearly independent from the decision to include the participant in the study. Participants will be treated with oral semaglutide (at least 4 weeks on maintenance dose) once daily with or without other oral antidiabetics (OADs) as per local label at the discretion of the treating physician.
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Semaglutide — Participants will receive oral semaglutide with or without other OADs as per local label at the discretion of the treating physician and is clearly independent from the decision to include the participant in the study.

SUMMARY:
The purpose of the study is to look at the change in blood sugar levels in people with type 2 diabetes who are using oral semaglutide and planning to fast during Ramadan. Participants will take oral semaglutide as prescribed by the study doctor. The study will last for about 5 months (20 weeks). Participants will be asked to complete a patient diary about how and when they take the oral semaglutide tablets. Participants will complete this diary during the study period as instructed by study doctor.

ELIGIBILITY:
Inclusion Criteria:

1. Signed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol)
2. The decision to initiate treatment with commercially available oral semaglutide has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician before and independently from the decision to include the patient in this study
3. Male or female, age above or equal to 18 years at the time of signing informed consent
4. Patients diagnosed with T2D who intend to fast during Ramadan
5. Patient should be on oral semaglutide (at least 4 weeks on maintenance dose) with or without other OADs
6. Available HbA1c value ≤ 30 days prior to the patient enrolment visit (V1) or HbA1c measurement taken in relation with the patient enrolment visit (V1) if in line with local clinical practice

Exclusion Criteria:

1. Previous participation in this study. Participation is defined as having given informed consent in this study
2. Participation in any clinical trial of an approved or non-approved investigational medicinal product within 30 days prior to the patient enrolment visit (V1) and throughout the duration of the study
3. Patients with type-1 diabetes and gestational diabetes
4. Patients who are pregnant or are planning to become pregnant during the conduct of the study
5. Patients who are breastfeeding
6. Patients on Insulin therapy within 2 weeks prior to enrolment
7. Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with T2D who intend to fast during Ramadan.
Sampling Method: Non-Probability Sample
Enrollment: 288 (Actual)
Dates: Start 2023-01-25 (Actual); Primary Completion 2023-07-09 (Actual); Study Completion 2023-07-09 (Actual)

PRIMARY OUTCOMES:
Change in glycated haemoglobin (HbA1c) | From participant enrolment visit (0 to 8 weeks before Ramadan) to end of follow-up visit (0 to 8 weeks after Ramadan)
  Percentage (%) of HbA1c.

SECONDARY OUTCOMES:
Relative change in body weight | From participant enrolment visit (0 to 8 weeks before Ramadan) to end of follow-up visit (0 to 8 weeks after Ramadan)
  Measured in percentage.
Absolute change in body weight | From participant enrolment visit (0 to 8 weeks before Ramadan) to End of follow-up visit (0 to 8 weeks after Ramadan)
  Measured in kilogram (kg).
Self-reported confirmed hypoglycaemic events | From participant enrolment visit (0 to 8 weeks before Ramadan) to end of follow-up visit (0 to 8 weeks after Ramadan)
  Measured in count of events.
Self-reported hyperglycaemic episodes requiring hospitalisation | From participant enrolment visit (0 to 8 weeks before Ramadan) to end of follow-up visit (0 to 8 weeks after Ramadan)
  Measured in count of episodes.
Number of participants reporting greater than or equal to (>= 1) severe hypoglycaemic events | From participant enrolment visit (0 to 8 weeks before Ramadan) to end of follow-up visit (0 to 8 weeks after Ramadan)
  Measured in count of participants.
Number of self-reported gastrointestinal (GI) side-effects | From participant enrolment visit (0 to 8 weeks before Ramadan) to end of follow-up visit (0 to 8 weeks after Ramadan)
  Measured in count of events.
Addition of new OAD or increased baseline OAD dose during the study period | At end of follow-up visit (0 to 8 weeks after Ramadan)
  Measured in count of participants (yes or no).
Removal of OAD or reduction of baseline OAD dose during the study period | At end of follow-up visit (0 to 8 weeks after Ramadan)
  Measured in count of participants (yes or no).
Increase in dose of oral semaglutide | From participant enrolment visit (0 to 8 weeks before Ramadan) to end of follow-up visit (0 to 8 weeks after Ramadan)
  Measured in count of participants (yes or no).
Decrease in dose of oral semaglutide | From participant enrolment visit (0 to 8 weeks before Ramadan) to end of follow-up visit (0 to 8 weeks after Ramadan)
  Measured in count of participants (yes or no).
Waiting time of at least 30 min after intake of oral semaglutide and before eating or drinking or taking any other oral medicinal product as per local label and as reported in patient diary | From participant enrolment visit (0 to 8 weeks before Ramadan) to end of follow-up visit (0 to 8 weeks after Ramadan)
  Measured in count of participants (yes or no).
Intake of oral semaglutide with up to 120 milliliter (mL) of water as reported in patient diary | From participant enrolment visit (0 to 8 weeks before Ramadan) to end of follow-up visit (0 to 8 weeks after Ramadan)
  Measured in count of participants (yes or no).
Timing of intake of oral semaglutide as reported in patient diary | From participant enrolment visit (0 to 8 weeks before Ramadan) to end of follow-up visit (0 to 8 weeks after Ramadan)
  Time before iftar (before iftar is before breaking the fast)/time before suhour (before suhour is before the last meal)/others.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (20):
- Kuwait (5):
  - KOC Hospital, Al Ahmadi
  - Al Seef Hospital, As Sālimīyah
  - Glycemia Clinic, As Sālimīyah
  - New Mowasat Hospital, As Sālimīyah
  - New Mowasat Clinics, Mangaf
- Saudi Arabia (8):
  - Almoosa Specialist Hospital, Ihsaa
  - Saudi German Hospital, Jeddah
  - Mouwasat Hospital Khobar, Khobar
  - Dr. Sulaiman Al Habib Medical Group- Olaya, Riyadh
  - Habib Medical Group, Riyadh
  - Al Hammadi, Riyadh
  - Dr. Sulaiman Al Habib Medical Group- Swedi, Riyadh
  - Dallah Hospital_Riyadh, Riyadh
- United Arab Emirates (7):
  - Thumbay Hospital Ajman, Ajman
  - Dubai Hospital, Dubai
  - Dubai Diabetes Center, Dubai
  - Al Garhoud Private Hospital, Dubai
  - Medcare Hospital, Dubai
  - NMC Specialty Hospital Dubai, Dubai
  - Oriana Hospital Sharjah, Sharjah city

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Hassanein M, Alawadi F, AlKadhim I, Aly H, Bajawi D, Cinar T, Dhanwal D, Jabbar A, Khader S, Khudadah K, Muzaffar T, Ngome M, Nafach J, Shaghouli A; O-SEMA-FAST Investigators. O-SEMA-FAST: A Prospective, Non-interventional Study Investigating Oral Semaglutide Use in Adults with Type 2 Diabetes Mellitus During Ramadan. Diabetes Ther. 2025 Apr;16(4):663-684. doi: 10.1007/s13300-025-01702-1. Epub 2025 Feb 28. PMID 40016571